CLINICAL TRIAL: NCT05455801
Title: Randomized Study on the Efficacy of Negative Pressure Wound Therapy (NPWT) in the Prevention of Surgical Site Complications
Brief Title: Study to Analyze the Surgical Site Infections in a Group of Patients Who Were Randomly Applied a Negative Pressure Therapy Dressing Versus Conventional Dressing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Central de Asturias (Other)
Responsible Party: Principal Investigator, María Moreno Gijon, Principal Investigator, Hospital Universitario Central de Asturias
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pNPWTHUCA
Record Dates: First submitted 2022-07-01; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Surgical Site Infection; Complication,Postoperative; Surgical Wound Infection; Surgical Complication
Keywords: surgical site infections; prophylaxis; negative pressure wound therapy; abdominal surgery
MeSH Terms: conditions — Surgical Wound Infection; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Randomly apply a negative pressure therapy dressing in the operating room to heal a surgical wound or a conventional dressing without negative pressure in those patients at high risk of presenting complications and surgical site infections
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- negative wound therapy group (Experimental): those who receive negative pressure therapy
  Interventions: Device: negative preassure wound therapy
- conventional dressing group (No Intervention): those patients who heal with conventional dressing, therefore negative pressure therapy is not applied

INTERVENTIONS:
Device: negative preassure wound therapy — wound treated with negative pressure therapy dressing
  Arms: negative wound therapy group

SUMMARY:
Surgical site complications generate a series of consequences that prolong hospital stay, increase interventions and procedures, and consequently considerably increase healthcare costs. Hence, the importance of studying measures to reduce these complications and the most feared of them is surgical site infection. The objective of the study is to analyze the complications of the surgical site in a group of participante with risk factors for developing them after undergone abdominal surgery in the period described.

DETAILED DESCRIPTION:
All non-consecutive participants operated on in a hospital were included, both those who, based on a protocol prepared by the investigators unit, were classified as having no risk of developing complications, low risk or high risk. Partfipants classified as low and high risk, after their consent to participate in the study, entered to form part of it. This participanta were classified before surgery according to the risk factors of themselves and of the procedure, and those at risk were randomized to treatment with a negative pressure therapy dressing or no treatment, and a cure was performed with a conventional dressing. The participants classified as not at risk of complications were not included in the study. In this way the investigators tried to analyze if the intervention with the negative pressure therapy dressing reduced the complications of the surgical site.The primary objective was to analyze the reduction of surgical site infections in participants treated with negative pressure therapy compared to those treated with conventional dressing. As secondary objectives the investigators proposed to measure other complications in both groups and the hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* patients with risk factors for developing surgical site complications
* undergo abdominal surgery
* consent of the patient to participate in the study

Exclusion Criteria:

* non-consent of the patient to participate in the study
* patients without risk of developing surgical site complications

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
surgical site complications | 30 days after surgery
  development of surgical site infection of wound seroma, skin dehiscence, wound necrosis

SECONDARY OUTCOMES:
length of hospital stay | 30 days
  days

CONTACTS AND LOCATIONS:
Locations (1):
- María Moreno Gijón, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bueno-Lledo J, Martinez-Hoed J, Pous-Serrano S. Negative pressure therapy in abdominal wall surgery. Cir Esp (Engl Ed). 2022 Aug;100(8):464-471. doi: 10.1016/j.cireng.2022.05.017. Epub 2022 May 16. PMID 35584763
- [Background] Wang XX, Xiang Y, Meng Y, Ma B, Hu XY, Tang HT, Ben DF, Xiao SC. [Clinical effects of negative pressure wound therapy in treating the poor healing of incisions after different abdominal operations]. Zhonghua Shao Shang Za Zhi. 2021 Nov 20;37(11):1054-1060. doi: 10.3760/cma.j.cn501120-20210518-00194. Chinese. PMID 34794257
- [Background] Mehdorn M, Jansen-Winkeln B. Modified Incisional Negative Pressure Wound Therapy Increases Seroma Evacuation: An Ex Vivo Model. Biomed Res Int. 2021 Oct 21;2021:5846724. doi: 10.1155/2021/5846724. eCollection 2021. PMID 34722767
- [Background] Ayuso SA, Elhage SA, Okorji LM, Kercher KW, Colavita PD, Heniford BT, Augenstein VA. Closed-Incision Negative Pressure Therapy Decreases Wound Morbidity in Open Abdominal Wall Reconstruction With Concomitant Panniculectomy. Ann Plast Surg. 2022 Apr 1;88(4):429-433. doi: 10.1097/SAP.0000000000002966. PMID 34670966
- [Background] Zhao AH, Kwok CHR, Jansen SJ. How to Prevent Surgical Site Infection in Vascular Surgery: A Review of the Evidence. Ann Vasc Surg. 2022 Jan;78:336-361. doi: 10.1016/j.avsg.2021.06.045. Epub 2021 Sep 17. PMID 34543711
- [Background] Gong S, Yang J, Lu T, Tian H, Huang Y, Song S, Lei C, Yang W, Yang K, Guo T. Incisional negative pressure wound therapy for clean-contaminated wounds in abdominal surgery: a systematic review and meta-analysis of randomized controlled trials. Expert Rev Gastroenterol Hepatol. 2021 Nov;15(11):1309-1318. doi: 10.1080/17474124.2021.1967143. Epub 2021 Aug 18. PMID 34384325
- [Background] Leuchter M, Hitzbleck M, Schafmayer C, Philipp M. Use of incisional preventive negative pressure wound therapy in open incisional hernia repair: Who benefits? Wound Repair Regen. 2021 Sep;29(5):759-765. doi: 10.1111/wrr.12948. Epub 2021 Jun 10. PMID 34110077
- [Background] Seaman AP, Sarac BA, ElHawary H, Janis JE. The effect of negative pressure wound therapy on surgical site occurrences in closed incision abdominal wall reconstructions: a retrospective single surgeon and institution study. Hernia. 2021 Dec;25(6):1549-1555. doi: 10.1007/s10029-021-02427-3. Epub 2021 May 19. PMID 34009506
- [Background] Almansa-Saura S, Lopez-Lopez V, Eshmuminov D, Schneider M, Castellanos-Escrig G, Rodriguez-Valiente M, Crespo MJ, von der Groeben M, Lehmann K, Robles-Campos R. Prophylactic Use of Negative Pressure Therapy in General Abdominal Surgery: A Systematic Review and Meta-Analysis. Surg Infect (Larchmt). 2021 Oct;22(8):854-863. doi: 10.1089/sur.2020.407. Epub 2021 Apr 12. PMID 33844934
- [Background] Roos E, Douissard J, Abbassi Z, Buchs NC, Toso C, Ris F, Meyer J. Prophylactic negative-pressure wound therapy for prevention of surgical site infection in abdominal surgery: a nationwide cross-sectional survey. Updates Surg. 2021 Oct;73(5):1983-1988. doi: 10.1007/s13304-021-01017-3. Epub 2021 Apr 10. PMID 33837948